CLINICAL TRIAL: NCT05397405
Title: A Prospective Observational Study on the Effect of Improving Blood Lipid Management on the Clinical Prognosis of Symptomatic Intracranial Atherosclerotic Stenosis（sICASBLM）
Brief Title: Improving Blood Lipid Management in Symptomatic Intracranial Atherosclerotic Stenosis on Clinical Outcome
Acronym: sICASBLM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sICASBLM
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Artery Stenosis
Keywords: symptomatic intracranial atherosclerotic stenosis; stroke; blood lipid management; PCSK9 inhibitors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Blood Lipid management with atorvastatin 20-40mg or rosuvastatin 10-20mg or simvastatin 20-40mg and PCSK9 inhibitors for 6-12 months
  Interventions: Drug: PCSK9 inhibitor
- Control group (No Intervention): Blood Lipid management with atorvastatin 20-40mg or rosuvastatin 10-20mg or simvastatin 20-40mg for 6-12 months

INTERVENTIONS:
Drug: PCSK9 inhibitor — The aim is to improve blood lipid management by using atorvastatin 20-40mg or rosuvastatin 10-20mg or simvastatin 20-40mg and PCSK9 inhibitors for 6-12 months
  Other Names: intensive blood lipid lowing
  Arms: Intervention group

SUMMARY:
sICASBLM is a prospective controlled trial, to asses the impact of improving blood lipid management on clinical outcome of moderate to severe symptomatic intracranial atherosclerotic stenosis patients (LDL-C>1.8mmol/L) without endovascular therapy.

DETAILED DESCRIPTION:
sICASBLM aims to determine the effectiveness of conventional lipid management combined with PCSK9 inhibitors compared to conventional lipid management (atorvastatin 20-40mg or rosuvastatin 10-20mg or simvastatin 20-40mg) in reducing the incidence of recurrent stroke in patients with moderate to severe symptomatic intracranial atherosclerotic stenosis (LDL-C>1.8mmol/L) without endovascular therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Symptomatic intracranial atherosclerotic stenosis of moderate to severe, did not receive intravenous thrombolysis, thrombectomy, stent implantation and other intravascular treatment
3. low density lipoprotein cholesterol > 70mg/dl (1.8mmol/L)
4. Receive 3T magnetic resonance angiography or multi-mode MR (high resolution is required), angiography can be included, and images for analysis can be obtained.
5. Lipid-lowering indications of statins
6. Signed an approved informed consents

Exclusion Criteria:

1. Contraindications to statins
2. There are contraindications to MRI examination or cannot accept MRI examination
3. Stenosis caused by vasculitis, arterial dissection and moyamoya disease
4. Patients with active bleeding or obvious bleeding tendency
5. Severe heart, lung, renal insufficiency, malignant tumor or other malignant diseases, and death is highly likely within 7 days; pregnancy or women who are lactating
6. Uncontrolled severe diabetes and hypertension
7. Other conditions inappropriate for inclusion judged by investigators

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke | 6 months-12 months
  the recurrent rate of clinical stroke

SECONDARY OUTCOMES:
Intracranial arterial | 6 months or 12 months
  Degree of change in intracranial arterial stenosis
Plaque changes | 6 months or 12 months
  Plaque volume and load changes
Vascular remodeling index | 6 months or 12 months
  Vascular remodeling index changes
Adverse events | 6 months or 12 months
  The incidence of muscle related events, allergic reactions, injection site reactions, bleeding events and other adverse events was assessed

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No